CLINICAL TRIAL: NCT01766076
Title: Use of Atorvastatin as Adjuvant Therapy Among Suboptimal Responders to Antiretroviral Therapy in an African Cohort of HAART-treated Adults: A Randomised Controlled Trial
Brief Title: Atorvastatin for HAART Suboptimal Responders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Makerere University (Other)
Collaborators: Vaccine and Gene Therapy Institute, Florida (Other)
Responsible Party: Principal Investigator, College of Health Sciences, Associate Professor, Makerere University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HS1258
Record Dates: First submitted 2012-12-10; First posted 2013-01-11 (Estimated); Results first posted 2015-05-21 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Acquired Immune Deficiency Syndrome Virus
Keywords: immune activation; antiretroviral therapy; atorvastatin; immune exhaustion; adults; Africa
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- atorvastatin, Lipitor® (Experimental): Intervention is be atorvastatin, Lipitor® (40mg) 2 tablets daily (as adjuvant to HAART) for 12 weeks.
  Peripheral blood mononuclear cells (PBMC) will be collected for immune activation assays using flowcytometry
  Interventions: Other: atorvastatin, Lipitor®; Drug: Placebo
- Placebo (Placebo Comparator): Intervention for the placebo comparator arm is Placebo 2 tablets daily for 12 weeks PBMC will be collected for immune activation assays using flowcytometry
  Interventions: Other: atorvastatin, Lipitor®; Drug: Placebo

INTERVENTIONS:
Other: atorvastatin, Lipitor® — PBMC collected for immune activation assays using flowcytometry
  Other Names: Lipitor®
Drug: Placebo — PBMC collected for immune activation assays using flowcytometry
  Other Names: atorvastatin placebo

SUMMARY:
We hypothesise that atorvastatin changes immune activation among HAART-treated adults with suboptimal cluster cell differentiation 4 (CD4) recovery by 25%

DETAILED DESCRIPTION:
The investigators have previously shown that up to 40% of HAART-treated adults have suboptimal CD4 recovery despite viral suppression. The investigators have also shown that immune activation and exhaustion are significantly higher among patients that do not exhibit satisfactory rise in CD4 counts despite viral suppression (suboptimal responders); when compared with their counterparts with viral suppression and satifactory CD4 count recovery (optimal responders). Given that atorvastatin changes immune activation in this pilot study, then larger studies can be done to understand its effect on CD4 count increase among suboptimal responders.

ELIGIBILITY:
List of inclusion Criteria: HIV-infected adults on antiretroviral therapy for at least 6 years with sustained viral suppression (viral load<400 copies), and CD4 increase below 300 cells (difference between current and baseline CD4 count).

List of exclusion Criteria: History of an opportunistic infection within the previous six months, Pregnancy, History of myositis, History of ingestion of lipid-lowering agents at the baseline visit, Use of therapeutic agents known to have substantial drug-drug interactions with statins, and individuals on PI-containing HAART

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-01; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Damalie Nakanjako, MD, PhD, Principal Investigator — Makerere University

REFERENCES:
- [Background] Ganesan A, Crum-Cianflone N, Higgins J, Qin J, Rehm C, Metcalf J, Brandt C, Vita J, Decker CF, Sklar P, Bavaro M, Tasker S, Follmann D, Maldarelli F. High dose atorvastatin decreases cellular markers of immune activation without affecting HIV-1 RNA levels: results of a double-blind randomized placebo controlled clinical trial. J Infect Dis. 2011 Mar 15;203(6):756-64. doi: 10.1093/infdis/jiq115. Epub 2011 Feb 15. PMID 21325137
- [Background] Nakanjako D, Ssewanyana I, Mayanja-Kizza H, Kiragga A, Colebunders R, Manabe YC, Nabatanzi R, Kamya MR, Cao H. High T-cell immune activation and immune exhaustion among individuals with suboptimal CD4 recovery after 4 years of antiretroviral therapy in an African cohort. BMC Infect Dis. 2011 Feb 8;11:43. doi: 10.1186/1471-2334-11-43. PMID 21299909

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 30 participants were recruited from the Infectious Diseases Institute research cohort (single site) and followed up for 12 weeks, 4 weeks wash out period and 12 weeks after cross over of treatment assignment
Pre-assignment Details: Participants were selected if they had sustained viral suppression for 7 years and CD4 increases below 300 cells/ul
Groups:
- Atorvastatin First, Then Placebo: Intervention is atorvastatin, Lipitor® (40mg) 2 tablets daily (as adjuvant to HAART) for 12 weeks.
  PBMC were collected for immune activation assays using flowcytometry
  'atorvastatin, Lipitor®': PBMC collected for immune activation assays using flowcytometry
- Placebo First, Then Atorvastatin: Intervention for the placebo comparator arm is Placebo 2 tablets daily for 12 weeks PBMC were collected for immune activation assays using flowcytometry
  Placebo: PBMC were collected for immune activation assays using flowcytometry
Period: Overall Study
Arm/Group | Atorvastatin First, Then Placebo | Placebo First, Then Atorvastatin
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Atorvastatin First, Then Placebo: Intervention is atorvastatin, Lipitor® (40mg) 2 tablets daily (as adjuvant to HAART) for 12 weeks.
  PBMC will be collected for immune activation assays using flowcytometry
  'atorvastatin, Lipitor®': PBMC were collected for immune activation assays using flowcytometry
- Placebo First, Then Atorvastatin: Intervention for the placebo comparator arm is Placebo 2 tablets daily for 12 weeks PBMC will be collected for immune activation assays using flowcytometry
  Placebo: PBMC were collected for immune activation assays using flowcytometry
- Total: Total of all reporting groups
Arm/Group | Atorvastatin First, Then Placebo | Placebo First, Then Atorvastatin | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 41 [40 to 50] | 47 [43 to 51] | 46 [40 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 8 | 5 | 13
Region of Enrollment [Number; unit: participants]
  Uganda | 15 | 15 | 30
CD4 T-cell activation [Median (Inter-Quartile Range); unit: percenatage of activated CD4 T-cells] | 4.2 [3.7 to 6.2] | 2.9 [2.9 to 5.0] | 4.2 [1.5 to 8.3]

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Immune Activation Levels After 12 Weeks of Atorvastatin 80mg Daily
Description: Immune activation was measured by co-expression of CD38 and HLADR on CD4 T-cells (CD4+CD38+HLADR+) Mean percentage change at 12 weeks was calculated
Time Frame: 12 weeks
Population: There was no cross-over or carry-over effect (the sequence did not matter), so we present data for 30 patients for their 12 weeks exposure to atorvastatin
Measure: Median (Inter-Quartile Range); unit: percentage change in activated T-cells
Groups:
- Atorvastatin: Intervention is be atorvastatin, Lipitor® (40mg) 2 tablets daily (as adjuvant to HAART) for 12 weeks.
  PBMC were collected for immune activation assays using flowcytometry
  'atorvastatin, Lipitor®': PBMC were collected for immune activation assays using flowcytometry
- Placebo: Intervention for the placebo comparator arm is Placebo 2 tablets daily for 12 weeks PBMC will be collected for immune activation assays using flowcytometry
  Placebo: PBMC were collected for immune activation assays using flowcytometry
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 30 | 30
percentage change in activated T-cells | 60 [50 to 68] | 21 [2 to 31]
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney); Mann Whitney test was used for nonparametric variables; Mean Difference (Final Values) = 28

ADVERSE EVENTS:
Time Frame: 12 weeks on study drug, 4 weeks wash out, then 12 weeks of placebo
Description: No serious adverse event reported
Groups:
- Atorvastatin First, Then Placebo: Intervention is atorvastatin, Lipitor® (40mg) 2 tablets daily (as adjuvant to HAART) for 12 weeks.
  PBMC were collected for immune activation assays using flowcytometry
  'atorvastatin, Lipitor®': PBMCwere collected for immune activation assays using flowcytometry
- Placebo First, Then Atorvastatin: Intervention for the placebo comparator arm is Placebo 2 tablets daily for 12 weeks PBMC wiere collected for immune activation assays using flowcytometry
  Placebo: PBMC were collected for immune activation assays using flowcytometry
Arm/Group | Atorvastatin First, Then Placebo | Placebo First, Then Atorvastatin
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 10/15 | 9/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin First, Then Placebo (N=15) | Placebo First, Then Atorvastatin (N=15)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) — 3 myalgias were reported in atorvastatin and placebo groups
Chest pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
headache (General disorders) | 1 (1) | 3 (3)
Joint pains (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
backache (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Abdominal pain (General disorders) | 0 | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
right forearm pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No